CLINICAL TRIAL: NCT04471649
Title: Clinical Course of COVID-19 in Patients With Rheumatoid Arthritis Treated With or Without Hydroxychloroquine: a Case-control Study
Brief Title: Hydroxy Chloroquine and Covid in RA Patients
Acronym: Covid-19
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Mohammed Hassan Abu-Zaid, Principal Investigator, Tanta University
Other Study IDs: 002
Record Dates: First submitted 2020-07-07; First posted 2020-07-15 (Actual); Last update posted 2020-09-09 (Actual); Status verified 2020-09

CONDITIONS: COVID
Keywords: Covid-19; Hydroxy chloroquine; Rheumatoid
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Experimental: Patient with rheumatoid arthritis using hydroxychloroquine as a part of their treatment regimen.
- Active Comparator: Patient with rheumatoid arthritis not using hydroxychloroquine as a part of their treatment regimen

SUMMARY:
evaluation of the clinical course of COVID-19 in a cohort of patients with rheumatoid arthritis treated with or without hydroxychloroquine.

DETAILED DESCRIPTION:
Study settings & sample:

This is an observational, retrospective -case-control, single-center study. This study will include patients who meet the inclusion criteria followed in the Department of Rheumatology and Rehabilitation, Tanta University Hospital, Tanta, Egypt.

Data will be taken from the medical records of patients with rheumatoid arthritis in the outpatient clinic of the Rheumatology and Rehabilitation Department, Tanta University Hospital, Tanta, Egypt. All patients will sign the informed consent form authorizing the collection of these data.

Group classification A) Patients with rheumatoid arthritis using hydroxychloroquine as a part of their treatment regimen.

b) Patients with rheumatoid arthritis not using hydroxychloroquine as a part of their treatment regimen.

Data will be collected and analyzed from patient medical records. It will include the following:

1. Epidemiologic, demographic, and clinical data.
2. Severity of rheumatoid arthritis.
3. Rheumatoid arthritis activity state using the Clinical Disease Activity Index
4. Dose and duration of hydroxychloroquine
5. Need for hospitalization, length of hospital stay, and ICU admission including the need for mechanical ventilation.
6. Duration from the start of symptoms until clinical cure.
7. Severity of COVID-19 disease according to the World Health Organization interim guidance
8. Prognosis.

Laboratory investigations and imaging:

1. Complete blood count.
2. Renal and liver function tests.
3. Random blood sugar.
4. Lactate dehydrogenase, D-dimer.
5. Serum ferritin, C-reactive protein,
6. Chest radiographs or CT scan

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with rheumatoid arthritis superinfected with Covid-19

Exclusion Criteria:

* Insufficient data are available in the medical record.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: To Evaluaye the clinical course of COVID-19 in a cohort of patients with rheumatoid arthritis treated with or without hydroxychloroquine:
  Data will be taken from the medical records of patients with rheumatoid arthritis in the outpatient clinic of the Rheumatology and Rehabilitation department, Tanta University hospital, Tanta, Egypt.
  A) Patient with rheumatoid arthritis using hydroxychloroquine as a part of their treatment regimen.
  b) Patient with rheumatoid arthritis not using hydroxychloroquine as a part of their treatment regimen.
  Primary Outcome Measures:
  1. Impact of hydroxychloroquine on the clinical course of Covid-19 in the hydroxychloroquine group compared to the non- hydroxychloroquine group.
  Data will be collected and analyzed from patient medical records.
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2020-06-15 (Actual); Primary Completion 2020-10 (Estimated); Study Completion 2020-11 (Estimated)

PRIMARY OUTCOMES:
Number of patients in need for hospitalization | through study completion an average 12 weeks
  Estimate number of patients in need for hospitalization
Length of hospitalization and ICU admission | through study completion an average 12 weeks
  Calculate the number of days that the patients stayed at the hospital and how many patients admitted to ICU
The need for mechanical ventilation | through study completion an average 12 weeks
  Calculate the number of patients who received mechanical ventilation
Severity of COVID-19 disease | through study completion an average 12 weeks
  WHO clinical management Covid19 interim guidance disease severity Algorithm

CONTACTS AND LOCATIONS:
Overall Officials: Asem Elfert, Prof, Study Chair — tanta university faculty of medicine
Locations (1):
- Tanta University Hospital, Tanta, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Cortegiani A, Ingoglia G, Ippolito M, Giarratano A, Einav S. A systematic review on the efficacy and safety of chloroquine for the treatment of COVID-19. J Crit Care. 2020 Jun;57:279-283. doi: 10.1016/j.jcrc.2020.03.005. Epub 2020 Mar 10. PMID 32173110